CLINICAL TRIAL: NCT00901498
Title: A Bioavailability Study of Four Experimental BMS-708163 Formulations Relative to Solubilized Capsule Formulation in Healthy Young Male Subjects
Brief Title: Relative Bioavailability Study of Four Experimental Formulations for Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CN156-004
Record Dates: First submitted 2009-05-05; First posted 2009-05-13 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer's Disease; Healthy
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Reference) (Experimental)
  Interventions: Drug: BMS-708163
- Treatment B (Active Comparator)
  Interventions: Drug: BMS-708163
- Treatment C (Active Comparator)
  Interventions: Drug: BMS-708163
- Treatment D (Active Comparator)
  Interventions: Drug: BMS-708163
- Treatment E (Active Comparator)
  Interventions: Drug: BMS-708163

INTERVENTIONS:
Drug: BMS-708163 — Oral, 25 mg Hard Gelatin Capsule, Size #2, 150 mg, Once per period of 3, 7 days between dosings. Will be compared with any 2 comparators.
  Arms: Treatment A (Reference)
Drug: BMS-708163 — Oral, 75 mg Tablet Formulation 1, 150 mg, Once per period of 3, 7 days between dosings
  Arms: Treatment B
Drug: BMS-708163 — Oral, 50 mg Hard Gelatin Capsule, Size #0, 150 mg, Once per period of 3, 7 days between dosings
  Arms: Treatment C
Drug: BMS-708163 — Oral, 75 mg Soft Gelatin Capsule, 150 mg, Once per period of 3, 7 days between dosings
  Arms: Treatment D
Drug: BMS-708163 — Oral, 75 mg Tablet Formulation 2, 150 mg, Once per period of 3, 7 days between dosings
  Arms: Treatment E

SUMMARY:
The purpose of this study is to assess the bioavailability of four experimental formulations relative to the current reference formulation used in the Phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy male subjects

Exclusion Criteria:

* Women

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To assess the bioavailability of 4 experimental formulations relative to the current reference formulation | Day 1, up to 3 weeks

SECONDARY OUTCOMES:
Safety: Adverse Events | Day 1, up to 3 weeks
Safety: Vital Signs | Screening, Day 1 and Day 4 of each period
Safety: ECGs | Screening, Day 1 of each period, up to 3 weeks
Safety: Clinical Lab Tests | Screening, Day -1 of each period, Day 1, up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mds Pharma Services (Us) Inc., Neptune City, New Jersey, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx